CLINICAL TRIAL: NCT04707404
Title: COMPREHENSIVE EVALUATION FOR CRANIOPLASTY WITH POLYETHERETHERKETONE AND TITANIUM IMPLANTS
Brief Title: Comparison of Cranioplasty With PEEK and Titanium
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Junfeng Feng, Prof., RenJi Hospital
Other Study IDs: RJCP2020
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Brain Injuries; Hematoma of Head; Skull Defect
Keywords: Cranioplasty; PEEK; Titanium; Outcomes; Complications; Subcutaneous effusion
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PEEK: Cranioplasty patients with PEEK.
  Interventions: Procedure: Cranioplasty
- Titanium: Cranioplasty patients with titanium mesh.
  Interventions: Procedure: Cranioplasty

INTERVENTIONS:
Procedure: Cranioplasty — The surgery implanted artificial material to repair the skull defect.

SUMMARY:
Decompressive craniectomy is suggested as an effective surgical intervention for patients with high intracranial pressure. Recently, various customized artificial materials are increasingly employed, e.g., titanium and polyetheretherketone (PEEK). The application of PEEK in cranioplasty is increasing, while its comprehensive evaluation in clinical practice is still insufficient, especially when comparing with the effects of titanium implant. We thus designed the study to evaluate the comprehensive effects of the cranioplasty with PEEK vs titanium.

DETAILED DESCRIPTION:
Decompressive craniectomy (DC) is suggested as an effective surgical intervention for patients with high intracranial pressure. For the skull defect after DC, cranioplasty could pro-vide protection, aesthetic and even functional improvements. The autologous bone flap (ABF) was once thought to be an optimal autograft for repairing [8]. While accumulated studies reported ABF related disadvantages. Recently, various customized artificial materials are increasingly employed, e.g., titanium and polyetheretherketone (PEEK).

Titanium is a widely applied metal material for cranioplasty, attribute to its high strength, bio-compatibility and comparatively low material cost. Currently, pre-operative three dimensional (3D) reconstruction of titanium brings a customized implant for optimal shaping effect. However, titanium implant is still confronted with complications of infection, implant exposure, etc.

PEEK is a novel polymer used to rebuild the personalized construction. Through the precise computational reconstruction of high-resolution computed tomography (CT) scanning, the customized PEEK could more accurately rebuild the complex cranial and maxillofacial structure. The application of this material in cranioplasty is increasing, while its comprehensive evaluation in clinical practice is still insufficient, especially when comparing with the effects of titanium implant.

We thus designed the study to evaluate the comprehensive effects of the cranioplasty with PEEK vs titanium. The data of the patients implanted PEEK or titanium in four years in our institute were retrospectively collected and evaluated, in respects of the general information of patients, postoperative complications, shaping effects, and psychosocial improvements, to display a comprehensive evaluation for these two implants.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent cranioplasty with PEEK or Titanium.
* Patients underwent cranioplasty and had complete data and 6-month follow-up records.

Exclusion Criteria:

* Patients underwent cranioplasty with other material or ABF.
* Patients had incomplete data or follow-up records.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients received cranioplasty with PEEK and titanium from December 2016 to July 2020 in Renji hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Complications | December 2016 to December 2020
  Postoperative complications including Incision infection, Subcutaneous infection, Postoperative hematoma, Subcutaneous effusion, New seizure, Implants exposure and Implants removal.

SECONDARY OUTCOMES:
Postoperative cranial symmetry | December 2016 to July 2020
  The postoperative cranial symmetry derived from the reconstruction of postoperative CT image.

OTHER OUTCOMES:
Postoperative improvement of GOSE score | December 2016 to Decemeber 2020
  The GOSE score in 6-month follow-up compared with the GOSE score in admission
Postoperative feelings | May 2017 to Decemeber 2020
  The subjective feelings for cranioplasty effect including 5 degrees of satisfaction and the Glasgow Benefit Inventory Score

IPD SHARING:
Plan to Share IPD: Undecided